CLINICAL TRIAL: NCT05296278
Title: Efficacy and Biomarker Explanation of IBI-323 Combined With Bevacizumab Plus Platinum Based Chemotherapy on ALK-Rearranged Non-Small Cell Lung Cancer Who Failed From First Line Alectinib
Brief Title: Efficacy and Biomarker Explanation of IBI-323 + Bevacizumab Plus Platinum Based Chemotherapy on ALK-Rearranged NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REVERSE
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): patients with only 3'ALK confirmed by NGS
  Interventions: Drug: IBI-323 combined with bevacizumab plus Platinum
- Cohort B (Experimental): patients with 3'ALK with retention of 5'ALK
  Interventions: Drug: IBI-323 combined with bevacizumab plus Platinum

INTERVENTIONS:
Drug: IBI-323 combined with bevacizumab plus Platinum — IBI-323 (30 mg/kg) ccombined with bevacizumab (15 mg/kg) plus platinum based chemotherapy ivgtt, every 21 days until disease progression

SUMMARY:
This study aimed to explore the efficacy and biomarker explanation of IBI-323 combined with bevacizumab plus platinum based chemotherapy on ALK-rearranged non-small cell lung cancer who failed from first line Alectinib.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent before implementing any trial-related procedures;
* Age ≥18 years old and ≤75 years old.
* No limit on the gender.
* Patients diagnosed with Lung Adenocarcinoma ALK-Rearranged Stage IIIA-IV by pathology.
* Patients who failed from first line Alectinib with stable brain metastasis included (Radiotherapy treated Oligo-metastasis).
* According to the Solid Tumor Efficacy Evaluation Criteria (RECIST V1.1), at least one lesion can be measured on imaging. Lesions located in the field of previous radiation therapy may be considered measurable if progression is demonstrated.
* ECOG score 0-1 points.

Exclusion Criteria:

* Patients with contraindication of chemotherapy Pregnant or breast feeding women.
* Participate in another interventional clinical study, unless participating in an observational (non-interventional) clinical study or in the survival follow-up phase of an interventional study.
* Participants are known to have had previous severe allergic reactions to other monoclonal antibodies or to any of the components of the IBI323 preparation, and severe allergies to bevacizumab, pemetrexed, cisplatin, and carboplatin.
* Previous systematic anti-tumor therapy for advanced non-squamous NSCLC other than ALK-TKI (including cytotoxic chemotherapy in combination with radiotherapy).
* Previous use of anti-PD-1 anti-PD-L1 anti-programmed death receptor ligand 2(PD-L2) or anti-cytotoxic T-lymphocyte-associated antigen 4(CTLA-4) drugs or any other drugs that act on T-cell co-stimulation or checkpoint pathways (such as OX40 CD137 LAG3, etc.).
* Radical radiation therapy within 28 days prior to the first dose, or palliative radiation therapy within 14 days prior to the first dose.
* Received ALK-TKI treatment within 2 weeks prior to the first administration of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects

SECONDARY OUTCOMES:
OS | 1 year
  Defined as the time from the start of treatment to the death of the subject due to any cause.
DCR | 1 year
  Disease control rates were assessed according to RECIST V1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China